CLINICAL TRIAL: NCT04787107
Title: The Effectiveness of a 10-minute Chair Massage Versus 10-minute Break to Reduce Psychological and Physical Stress in Healthcare Workers
Brief Title: Effectiveness of 10-minute Chair Massage Versus 10-minute Break to Reduce Stress and Improve Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Tami Underhill (Unknown)
Responsible Party: Principal Investigator, Sarah A. Evans, Director of Nursing Research, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0186
Record Dates: First submitted 2021-02-23; First posted 2021-03-08 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Stress, Psychological; Fatigue; Quality of Life
MeSH Terms: conditions — Stress, Psychological; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 Minute Chair Massage (Experimental): Chair massage for 10 minutes once a week for 5 weeks
  Interventions: Device: Mechanical Chair Massage
- 10 Minute Scheduled Break (Experimental): Scheduled 10-minute break once a week for 5 weeks
  Interventions: Device: Mechanical Chair Massage

INTERVENTIONS:
Device: Mechanical Chair Massage — Healthcare staff will be placed into either massage or break intervention
  Other Names: Schedule Break

SUMMARY:
The purpose of this study is to examine the effectiveness of 10-minute chair massage therapy in comparison to a scheduled 10-minute break to evaluate the impact on perceived quality of life, heart rate, blood pressure, and pain scale in healthcare workers.

DETAILED DESCRIPTION:
The primary purpose of this study is to provide cost-effective interventions for nursing personnel aimed at reducing fatigue and stress within their work environment while improving their overall quality of life. Studies have demonstrated that stress management resources and overall engagement of staff lead to quality outcomes for both staff and patients. There is limited research that examines interventions that can reduce stress perception in nursing. This study will examine the physical and psychological impact of 10-minute massage therapy in comparison to a 10-minute scheduled break weekly over a period of 5 weeks. If the outcomes of the study indicate that either massage therapy or scheduled breaks are an effective intervention for management of stressful situations and improving quality of life, the overall goal would be to create relaxation rooms on more nursing units that allow staff to engage in massage therapy or scheduled rest sessions to reduce stressful work situations.

Studies have indicated that healthcare workers experience high levels of work-related stress that include individual, social, occupational and environmental factors. Unrelieved or mismanaged stressors contribute to a variety of health-related consequences including disturbances in the digestive system, headaches, sleep disturbances, hypertension, fatigue and psychological issues, including anxiety. Massage therapy and scheduled breaks have been identified as potential interventions to mitigate or reduce stress. The use of mechanical massage has been shown to mimic the effects of traditional physical massage in terms of reducing stress and anxiety of the end-users. Mechanical massages have an advantage over physical massages since they are more cost-effective, can be used when convenient, and within a controlled environment. The literature supports that massage therapy can have an impact on reducing stress, anxiety, depression, and pain, while enhancing an individual's immune function, relaxation, and overall well-being. Studies have also indicated that nurses often lack opportunities to take breaks during their scheduled shifts. In many instances, staff sacrifice their breaks in order to fulfill patient-care duties. This study will compare both massage therapy and scheduled breaks to examine the overall impact on healthcare workers.

The COVID-19 pandemic has increased workplace stressors for healthcare workers; however, there is limited evidence to support successful interventions to manage these stressors.

ELIGIBILITY:
Inclusion Criteria:

* Health care professional assigned work duties on designed unit
* Men and women able age 18-84 able to give informed consent
* Able to speak and understand English

Exclusion Criteria:

* Individuals that decline to participate in the study
* Individuals currently on work restrictions
* Recent head, neck, shoulder or back surgeries

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Professional Quality of Life Scores | 5 weeks
  The change in professional quality of life scores will be compared pre trial and post at completion of 5 weeks

SECONDARY OUTCOMES:
Change in Heart Rate of 2-arms | 5 weeks
  Participants will record heart rate pre and post intervention for each session and these measures will be examined for decrease in heartrate and compared amongst both arms
Change in Blood Pressure of 2-arms | 5 weeks
  Participants will record blood pressure pre and post intervention for each session and these measures will be examined for decrease in blood pressure and compared amongst both arms
Change in Self-reported level of pain on scale of 0-10 | 5 weeks
  Participants will record self-reported pain level pre and post intervention for each session and these measures will be examined for decrease in level of pain and compared amongst both arms. Participants will use the Geisinger Pain Scale, 0 indicates no pain, 10 would indicate severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No